CLINICAL TRIAL: NCT01619527
Title: A Single-Dose, Open-Label, 3-Panel, Randomized, Pivotal Crossover Study to Assess the Bioequivalence of Darunavir When Co-Administrated With Cobicistat as Either a Fixed Dose Combination Tablet (G006) or as Single Agents Under Fed and Fasted Conditions in Healthy Subjects
Brief Title: A Study to Assess the Bioequivalence of Darunavir When Co-Administrated With Cobicistat Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100699; TMC114IFD1003 (Other: Janssen R&D Ireland); 2012-000273-23 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Darunavir; Cobicistat; Bioequivalence; Fixed dose combination; Pharmacokinetics; Human immunodeficiency virus; Protease inhibitor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Experimental): Single-dose co-administration of 800 mg darunavir and 150 mg cobicistat as single agents (under fasted condition)
  Interventions: Drug: darunavir; Drug: cobicistat
- Treatment B (Experimental): Single-dose co-administration of the fixed dose combination darunavir/cobicistat (800/150-mg) (under fasted condition).
  Interventions: Drug: darunavir; Drug: cobicistat
- Treatment C (Experimental): Single-dose co-administration of 800 mg darunavir and 150 mg cobicistat as single agents (under fed condition - standardized breakfast).
  Interventions: Drug: darunavir; Drug: cobicistat
- Treatment D (Experimental): Single-dose co-administration of the fixed dose combination darunavir/cobicistat (800/150-mg) (under fed condition - standardized breakfast).
  Interventions: Drug: darunavir; Drug: cobicistat
- Treatment E (Experimental): Single-dose co-administration of the fixed dose combination darunavir/cobicistat 800/150-mg (under fasted condition).
  Interventions: Drug: darunavir; Drug: cobicistat
- Treatment F (Experimental): Single-dose co-administration of the fixed dose combination darunavir/cobicistat (800/150-mg) (under fed condition - high-fat breakfast).
  Interventions: Drug: darunavir; Drug: cobicistat

INTERVENTIONS:
Drug: darunavir — Type=exact number, unit=mg, number=400, form=tablet, route=oral. Two tablets as a single dose or a tablet in combination with cobicistat
Drug: cobicistat — Type=exact number, unit=mg, number=150, form=tablet, route=oral. One tablet as a single dose or a tablet in combination with darunavir

SUMMARY:
The purpose of this study is to evaluate the single-dose pharmacokinetics and bioequivalence of darunavir 800 mg when administered as a fixed dose combination relative to 2 x 400 mg tablets of the commercial tablet formulation, in the presence of 150 mg cobicistat, (under fed and fasted conditions) in healthy participants.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), open-label (all people know the identity of the intervention), 3-panel, single-center, single-dose, crossover (method used to switch patients from one treatment arm to another in a clinical trial) study in 134 healthy adult participants. The study consists of 3 phases including a screening phase of approximately 3 weeks (Days -21 to -1) followed by an open-label treatment phase consisting of 3 panels with 2 single-dose treatment sessions of 5 days each (Days -1 to 4) separated by a washout period of at least 7 days, and a follow-up period occurring 7 to 10 days after last intake of study drugs. The study consists of 3 panels. In each panel participants will be randomly be assigned to 1 of 2 treatment sequences (AB or BA for Panel 1; CD or DC for Panel 2; and EF or FE for Panel 3). Participants will receive either single-dose darunavir 800 mg as 2 x 400 mg tablets and cobicistat 150 mg tablet or single-dose darunavir/cobicistat 800/150 mg as tablet in each panel (under fed and fasted conditions).

ELIGIBILITY:
Inclusion Criteria:

* Participant should be healthy on the basis of physical examination, medical history, vital signs, and electrocardiogram and clinical laboratory tests performed at screening
* Have a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.5 to 30.0 kg/m2, extremes included
* Men and women must agree to use a highly effective method of birth control

Exclusion Criteria:

* Has a positive HIV-1 or HIV-2 test at screening
* Has a Hepatitis A, B or C infection (confirmed by hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody, respectively) at screening
* Has any history of renal insufficiency
* Has a history of significant skin reactions or any history of allergies to drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Comparison of maximum plasma analyte concentration (Cmax) of darunavir as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg) | Up to 27 Days
  The pharmacokinetic parameter (Cmax) of darunavir will be compared as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg).
Comparison of last observed measurable analyte concentration (Clast) of darunavir as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg) | Up to 27 Days
  The pharmacokinetic parameter (Clast) of darunavir will be compared as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg).
Comparison of actual sampling time to reach the maximum plasma analyte concentration (tmax) of darunavir as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg) | Up to 27 Days
  The pharmacokinetic parameter (tmax) of darunavir will be compared as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg) for assessment of bioequivalance.
Area under curve from time of administration up to the last time point with a measurable plasma analyte concentration (AUClast) of darunavir as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg) | Up to 27 Days
  The pharmacokinetic parameter (AUClast) of darunavir will be compared as a fixed dose combination relative to 2 tablets of darunavir (400 mg), in the presence of cobicistat (150 mg).

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerabilty | Up to 27 Days
  Safety and tolerability of darunavir/cobicistat co-administration in healthy participants will be assessed by number of participants with adverse events.
Evaluation of plasma pharmacokinetics of cobicistat with darunavir when both administered as a fixed dose combination tablet | Up to 27 Days
  Plasma pharmacokinetics of cobicistat with darunavir when both administered as a fixed dose combination tablet under fed conditions in healthy participants will be evaluated.
Evaluation of plasma pharmacokinetics of cobicistat with darunavir when both administered as a single agents | Up to 27 Days
  Plasma pharmacokinetics of cobicistat with darunavir when both administered as a single agents under fed conditions in healthy participants will be evaluated.
Evaluation of plasma pharmacokinetics of cobicistat with darunavir when both administered as a fixed dose combination tablet | Up to 27 Days
  Plasma pharmacokinetics of cobicistat with darunavir when both administered as a fixed dose combination tablet under fasted conditions in healthy participants will be evaluated.
Evaluation of plasma pharmacokinetics of cobicistat with darunavir when both administered as a single agents | Up to 27 Days
  Plasma pharmacokinetics of cobicistat with darunavir when both administered as a single agents under fasted conditions in healthy participants will be evaluated
Evaluation of effect of a high-fat meal on darunavir and cobicistat pharmacokinetics relative to the fasted state | Up to 27 Days
  Effects of a high-fat meal on darunavir and cobicistat pharmacokinetics relative to the fasted state will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Merksem, Belgium